CLINICAL TRIAL: NCT06636643
Title: The Effect of Bone Marrow Stem Cells Harvested from the Iliac Crest Versus Mandibular Ramus in Alveolar Cleft Regeneration
Status: Completed | Type: Observational
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Doaa Selim, Doaa selim, Faculty of Dental Medicine for Girls
Other Study IDs: Al azhar university
Record Dates: First submitted 2024-10-07; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Cleft Lip and Palate
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- received Autologous (BMMSCs) harvested from the mandibular ramus and seeded on a collagen sponge in: received Autologous (BMMSCs) harvested from the lilac crest and seeded on a collagen sponge in combination with nanohydroxyapatite.

SUMMARY:
This comparative and prospective study was conducted on 10 patients with alveolar cleft defects. Patients with alveolar cleft defects were randomly selected and randomly divided into two equal groups: Group A: received Autologous (BMMSCs) harvested from the mandibular ramus and seeded on a collagen sponge in combination with nanohydroxyapatite. Group B: received Autologous (BMMSCs) harvested from the lilac crest and seeded on a collagen sponge in combination with nanohydroxyapatite.

DETAILED DESCRIPTION:
The utilization of Mandibular Ramus-derived BMSCs presents a groundbreaking advancement in maxillofacial reconstruction. This approach offers numerous advantages, including reduced surgical complications, improved precision and localization, higher osteogenic potential, and lower risks of graft rejection. Moreover, the combination of BMMNCs, nanohydroxyapatite, and PRF extracted from the mandible proves to be a viable alternative to traditional iliac crest grafting, promoting effective bone regeneration in alveolar cleft defects. By adopting this novel technique and harvesting site, It can can optimize surgical interventions, paving the way for enhanced standards of care and improving the quality of life for patients with maxillofacial challenges

ELIGIBILITY:
Inclusion Criteria:

* patient aged 8-15 years, not received any surgery for alveolar cleft defect, non-syndromic unilateral alveolar cleft with or without cleft palate, good oral hygiene and good compliance with the plaque-control instructions, medically fit for major surgical oral procedure.

Exclusion Criteria:

* pre-existing infection at the cleft site, patients with systemic diseases may affect bone healing.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with alveolar cleft defects randomly divided into two equal groups: Group A: received Autologous Bone Marrow Mesenchymal Stem Cells (BMMSCs) harvested from the mandibular ramus and seeded on a collagen sponge in combination with nanohydroxyapatite. Group B: received Autologous Bone Marrow Mesenchymal Stem Cells (BMMSCs) harvested from the lilac crest and seeded on a collagen sponge in combination with nanohydroxyapatite
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
The utilization of Mandibular Ramus-derived BMSCs presents a groundbreaking advancement in maxillofacial reconstruction. This approach offers numerous advantages, including reduced surgical complications | 6 months
  Based on the given data, there is a significant difference the volume reduction was significantly different between both groups being better in group A compared to group B (P=0.047). Whereas there was an insignificant difference between both groups regarding the preoperative and postoperative volume area.

CONTACTS AND LOCATIONS:
Locations (1):
- Al azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26973535/